CLINICAL TRIAL: NCT04208867
Title: Strengthening People-centered Accessibility, Respect, and Quality for Reproductive Health Services in Uttar Pradesh, India, Phase 1
Brief Title: Quality Improvement Project for Reproductive Health Services in India, Phase 1
Acronym: SPARQ_QII1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Population Services International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-18008_IndiaQI1
Record Dates: First submitted 2019-12-18; First posted 2019-12-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Maternal Health; Delivery; Reproductive Health
Keywords: Maternal Health; Delivery; Person-centered Care; India; Family Planning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention - Women (Experimental): Women who receive MH services from a facility participating in the QI collaborative to improve PCC
  Interventions: Behavioral: QI Collaborative
- Control - Women (No Intervention): Women who receive MH services from a facility not participating in the QI collaborative to improve PCC
- Intervention - Provider (Experimental): Provider working at a facility participating in the QI collaborative to improve PCC
  Interventions: Behavioral: QI Collaborative
- Control - Provider (No Intervention): Provider working at a facility not participating in the QI collaborative to improve PCC

INTERVENTIONS:
Behavioral: QI Collaborative — Facilities that participated in a QI collaborative to improve PCC for MH services
  Arms: Intervention - Provider; Intervention - Women

SUMMARY:
Evaluation of a quality improvement (QI) collaborative aimed at improving person-centered care (PCC) for reproductive health (RH) services.

DETAILED DESCRIPTION:
Evaluation of a quality improvement (QI) collaborative in public facilities in Uttar Pradesh, India aimed at improving person-centered care (PCC) for reproductive health (RH) services.

ELIGIBILITY:
Inclusion Criteria for Women:

* Women aged 18-49
* Agree/consent to participate
* Delivered a baby at the facility within 7 days (or adopted a family planning method at time of visit (baseline only, not part of intervention))

Exclusion Criteria for Women:

* Not a women aged 18-49
* Did not agree/consent to participate
* Did not deliver a baby at the facility within 7 days (or adopted a family planning method at time of visit (baseline only, not part of intervention))

Inclusion Criteria for Providers:

* Agreed/consented to participate
* Staff at facility

Exclusion Criteria for Provider:

* Did not agree/consent to participate
* Not Staff at facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2989 (Actual)
Dates: Start 2016-09-16 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2018-12-06 (Actual)

PRIMARY OUTCOMES:
Person Centered Maternal Health Scale Score | Baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-100; higher the score the better the experience of care
Person Centered Maternal Health Scale Score | 2-weeks post basline
  Survey conducted with women: self report of experiences of care. Possible range 0-100; higher the score the better the experience of care
Person Centered Maternal Health Scale Score | 4 weeks post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-100; higher the score the better the experience of care
Person Centered Maternal Health Scale Score | 10 weeks post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-100; higher the score the better the experience of care
Person Centered Maternal Health Scale Score | About 12 months post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-100; higher the score the better the experience of care
Person Centered Maternal Health Scale Score | About 14 months post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-100; higher the score the better the experience of care
Person Centered Maternal Health Scale Score | about 24 months after baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-100; higher the score the better the experience of care
Person Centered Maternal Health Scale Score | About 24.5 months post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-100; higher the score the better the experience of care
Person Centered Maternal Health Scale Score | 25 months post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-100; higher the score the better the experience of care
Person Centered Maternal Health Scale Score | 26.5 months past baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-100; higher the score the better the experience of care
Person Centered Family Planning Scale Score | Baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-43; higher the score the better the experience of care
Person Centered Family Planning Scale Score | 4 weeks post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-43; higher the score the better the experience of care
Person Centered Family Planning Scale Score | 10 weeks post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-43; higher the score the better the experience of care
Attitude toward Person-Centered Care | About 12 months post baseline
  Survey and in-depth interviews conducted with providers; perceptions of person-centered care
Attitude toward Person-Centered Care | About 24 months post baseline
  Survey and in-depth interviews conducted with providers; perceptions of person-centered care

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Montagu, DrPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Population Services International, Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Montagu D, Giessler K, Nakphong MK, Green C, Roy KP, Sahu AB, Sharma K, Sudhinarset M. A comparison of intensive vs. light-touch quality improvement interventions for maternal health in Uttar Pradesh, India. BMC Health Serv Res. 2020 Dec 4;20(1):1121. doi: 10.1186/s12913-020-05960-6. PMID 33276773